CLINICAL TRIAL: NCT03905499
Title: Can Robot Assited Physical Therapy Affect Pseudoparalysis in Patients Treated for Massive Rotator Cuff Tear? A Feasibility Study
Brief Title: Robot Assisted Physical Therapy for Pseudoparalysis in Massive Rotator Cuff Tear
Status: Available | Type: Expanded Access
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Other Study IDs: OE-0067 (RC-Pseudoparalysis)
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Pseudoparalysis Due to Massive Rotator Cuff Tear
Keywords: Massive rotator cuff tear; Pseudoparalysis; Robotic mediated therapy

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Device: Robotic assisted therapy with MJS (multi joint system) Tecnobody — The intervention will include 18 30-minutes trainings evenly distributed over a time period of 6 weeks and will be administered by the same two physiotherapists at the Schulthess clinic based on the standardized protocol
Other: Usual Care — Patients randomized in the usual care will receive standard of care treatment without receiving any active intervention

SUMMARY:
The primary objective of this study is to assess the efficacy of a robot assisted therapy in a clinical setting and its potential benefit for patients with rotator cuff tear associated with pseudoparalysis. eighty patients with clinical signs of pseudoparalysis will be recruited through doctors and physical therapists based on eligibility criteria. After completing the baseline assessments, patients will be randomized into the robot-assisted physical therapy intervention or control comparison group. Enrolled patients will conduct a specific trainings program with the MJS Tecnobody (Multi Joint System 614P Tecnobody Srl, IT) three times a week over a period of six weeks. Feasibility assessment will be performed six and twelve weeks after baseline and secondary outcomes (Oxford shoulder score, subjective shoulder value, pain level during activity of daily living, active shoulder flexion and abduction and quality of life EQ-5D-5L) will be assessed at baseline, six and twelve weeks post intervention.

DETAILED DESCRIPTION:
Rotator cuff tears are a common disorder in chronic shoulder pain. Common Complaints are pain, loss of range of motion and loss of strength. 20% of all tears are massive, in re-ruptures even 80%, with at least two tendons involved and this could lead to pseudoparalysis. The recommendation for the initial treatment is non-operative with physical therapy although people often receive a shoulder endoprosthesis. Robotic mediated therapy in patients with neurological disorders is already common, in rotator cuff tears it is less frequent and evidence is rare though. Therefore, the primary objective of this study is to evaluate the feasibility of a robotic mediated therapy in a clinical setting, in terms of satisfaction, compliance and tolerance, and its potential benefit for patients with rotator cuff tear associated with pseudoparalysis.

Eighty patients with clinical signs of pseudoparalysis will be recruited in the Schulthess clinic in Zurich through doctors and physical therapists of the shoulder and elbow surgery department based on eligibility criteria. Eligible patient will be enclosed after signing the informed consent. The patients will attend a specific trainings program with the MJS Tecnobody (Multi Joint System 614P Tecnobody Srl, IT) three times a week over a period of six weeks. The training is guided by a specialised physical therapist and the trainings program is developed by physical therapists and doctors of the Schulthess clinic based on current literature. Feasibility assessment will be performed six and twelve weeks after baseline and secondary outcomes (Oxford shoulder score, subjective shoulder value, pain level during activity of daily living, active shoulder flexion and abduction and quality of life EQ-5D-5L) will be assessed at baseline, six and twelve weeks post intervention. Primary analysis will be descriptive and secondary analysis will be analyzed with a univariate paired non-parametric analysis. All statistical tests will be two-sided and the level of significance will be set at p < 0.05. We will follow a repeated measures analysis to investigate changes in the outcomes variables across time. This approach allows for the examination of within-subject differences, making it particularly useful in studying interventions or treatments where individuals serve as their own control.

ELIGIBILITY:
Inclusion Criteria:

* Active flexion <45°
* Massive, irreparable, atraumatic RC tear at least two tendons
* Almost full passive ROM glenohumeral (140-180°)
* Fatty infiltration of the muscle Goutallier grade III or IV
* Persistent loss of active ROM after injection
* Ability to speak and understand German or English

Exclusion Criteria:

* Neurological disease
* Clinical diagnosis of rheumatoid arthritis, glenohumeral osteoarthritis, periarthritis and necrosis
* RC repair in the previous two years
* Acute fracture
* Acute traumatic RC tear
* Capsular shoulder stiffness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Markus Scheibel, Dr, Principal Investigator — Schulthess Klinik
Locations (1):
- Schulthess Klinik, Zurich, Canton of Zurich, Switzerland